CLINICAL TRIAL: NCT01895023
Title: Dexmedetomidine Versus Midazolam Premedication on Emergence Agitation After Strabismus Surgery in Children
Brief Title: Effects of Dexmedetomidine Premedication on Emergence Agitation After Strabismus Surgery in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yao Yusheng (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor-Investigator, Yao Yusheng, Dr., Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FujianPH-TRC-130615
Record Dates: First submitted 2013-06-28; First posted 2013-07-10 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Inhalational Anesthetics Adverse Reaction; Delirium on Emergence; Strabismus Following Ocular Surgery
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Midazolam; GABA Modulators; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexmedetomidine group (Experimental): The dexmedetomidine group received intranasal dexmedetomidine 2mcg/kg premedication 45 min and oral saline 30 min before induction of anaesthesia
  Interventions: Drug: Dexmedetomidine
- Midazolam group (Active Comparator): The midazolam group received intranasal saline 45 min and oral midazolam 0.5 mg/kg 30 min before induction of anaesthesia.
  Interventions: Drug: Midazolam
- Placebo Group (Placebo Comparator): The Placebo group received intranasal saline premedication 45 min and oral saline 30 min before induction of anaesthesia
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — The dexmedetomidine group received intranasal dexmedetomidine 2mcg/kg premedication 45 min before induction of anaesthesia.
  Other Names: alpha2-adrenoceptor agonist
  Arms: Dexmedetomidine group
Drug: Midazolam — The midazolam group oral midazolam 0.5 mg/kg 30 min before induction of anaesthesia.
  Other Names: GABA modulators
  Arms: Midazolam group
Drug: Saline — The Placebo group received intranasal saline premedication 45 min and oral saline 30 min before induction of anaesthesia
  Other Names: sodium chloride injection (0.9%Nacl)
  Arms: Placebo Group

SUMMARY:
Sevoflurane is frequently used for pediatric anesthesia because it has low pungency and rapid onset and offset of action.The reported incidence of emergence agitation (EA) following sevoflurane anesthesia varies from 10-80%. Despite its spontaneous resolution, EA is still considered as a potentially serious complication because of the risks of self-injury, and because of the stress caused to both caregivers and families.

Dexmedetomidine, an Alpha2-adrenoceptor agonist with sedative, analgesic, and anxiolytic actions, has been used in pediatric populations.Several prospective clinical trials in children have shown that dexmedetomidine significantly reduces the incidence of EA prior to recovery from sevoflurane anesthesia. However, the effect of dexmedetomidine premedication on emergence agitation has not been fully evaluated. The purpose of the present study was to verify the hypothesis that intranasal premedication with dexmedetomidine is effective in reducing emergence agitation after sevoflurane anaesthesia.

DETAILED DESCRIPTION:
Emergence agitation was assessed using the Pediatric Anesthesia Emergence Delirium (PAED) scale.The PAED scale contains five items (eye contact, purposefulness of actions,awareness of surroundings, restlessness and consolability), each scored on a 0 to 4 scale, for a maximum of 20 points.

A perfectly calm child scores 0 and extreme agitation corresponds to 20 points. The peak EA score was recorded. Agitation scores < 10 were interpreted as an absence of agitation, scores>= 10 were regarded as presence of agitation.

ELIGIBILITY:
Inclusion Criteria:

* aged2-6 yr, with American Society of Anesthesiologists physical status I or II, scheduled to undergo strabismus surgery during general anesthesia

Exclusion Criteria:

* mental disease, neurologic disease, treatment with sedatives, full stomach, or indication for rapid sequence induction.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Emergence agitation | participants will be followed for the duration of PACU stay, an expected average of 1 hour
  Emergence agitation was assessed using the Pediatric Anesthesia Emergence Delirium (PAED) scale.The PEAD scale contains five items (eye contact, purposefulness of actions,awareness of surroundings, restlessness and consolability), each scored on a 0 to 4 scale, for a maximum of 20 points.
  A perfectly calm child scores 0 and extreme agitation corresponds to 20 points. The peak EA score was recorded. scores>= 10 were regarded as presence of agitation.

SECONDARY OUTCOMES:
Postoperative vomiting | up to 24 hours
  Postoperative vomiting was assessed using a numeric rank score, where 0 = no vomiting,1 = vomited once, and 2 = vomited twice or more

OTHER OUTCOMES:
Children's pain | participants will be followed for the duration of PACU stay, an expected average of 1 hour
  A Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) was used to measure five categories of pain related behaviour, each scored from 0, 1 or 2, for a maximum score of 10.
Time of emergence | up to 1 hour
  the time to the first response to a simple verbal command
Duration of PACU stay | participants will be followed for the duration of PACU stay, an expected average of 1 hour
  The subject was discharged from the PACU when they met the institutional guidelines of level of consciousness and comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Yusheng Yao, M.D., Principal Investigator — Fujian Provincial Hospital
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Yao Y, Sun Y, Lin J, Chen W, Lin Y, Zheng X. Intranasal dexmedetomidine versus oral midazolam premedication to prevent emergence delirium in children undergoing strabismus surgery: A randomised controlled trial. Eur J Anaesthesiol. 2020 Dec;37(12):1143-1149. doi: 10.1097/EJA.0000000000001270. PMID 32976205